CLINICAL TRIAL: NCT03469700
Title: General Anesthesia vs Paravertebral Block With General Anesthesia For Post-Operative Pain Post Laparoscopic Sleeve Gastrectomy
Brief Title: General Anesthesia vs Paravertebral Block With General Anesthesia For Laparoscopic Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Saleh Kanawati, Anesthesiologist, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 15218
Record Dates: First submitted 2018-03-03; First posted 2018-03-19 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GA+PVB (Experimental): Patients will receive general anesthesia with paravertebral block
  Interventions: Other: general anesthesia; Other: Paravertebral block
- GA+placebo PVB (Active Comparator): Patients will receive general anesthesia with placebo block
  Interventions: Other: general anesthesia; Other: Placebo PVB

INTERVENTIONS:
Other: general anesthesia — Induction of general anesthesia will be performed followed by endotracheal intubation. General anesthesia is induced with 0.5-1 μg/kg fentanyl, 1.5-2 mg/kg propofol and 1-2 mg midazolam. Then, endotracheal intubation is facilitated by 0.15 mg/kg nimbex. Anesthesia is maintained by 1-1.5% sevoflurane, 0.5 μg/kg/h fentanyl, 0.6 mg/kg/h rocuronium, 60% nitrous oxide and 40% oxygen with Ultiva (Remifentanyl) 0.1-0.2 μg/kg/hr
Other: Paravertebral block — Bilateral paravertebral block guided by a nerve stimulator will be performed by injecting local anesthetic mixture from levels T11 to T6. Each 20 ml of the mixture will contain: 6 ml lidocaine 2%; 6 ml lidocaine 2% with adrenaline 5 μg /ml; 5 ml bupivacaine 0.5%; 50μg fentanyl (1 ml); and 2 ml saline 0.9%
  Arms: GA+PVB
Other: Placebo PVB — Placebo bilateral paravertebral block guided by a nerve stimulator will be performed by injecting normal saline from levels T11 to T6.
  Arms: GA+placebo PVB

SUMMARY:
The incidence of obesity is steadily rising. Laparoscopic sleeve gastrectomy (LSG) is an innovative approach to the surgical management of morbid obesity.

We will be discussing the effect of adding paravertebral block (PVB) in addition to general anesthesia (GA) vs. GA alone for post operative pain after laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind controlled clinical trial. Written informed consent will be obtained from patients. Patients will be randomly assigned using the sealed envelope technique into 2 equal groups: Group 1 will be patients who receive general anesthesia with paravertebral block, whereas group 2 will be patients who receive general anesthesia with placebo block.

ELIGIBILITY:
Inclusion Criteria:

* Patients with body mass index (BMI) greater than or equal to 30
* American Society of Anesthesiologist (ASA) score greater than or equal to 2
* Undergoing laparoscopic gastric sleeve surgeries

Exclusion Criteria:

* Patients with ASA score less than 2 and greater than 4
* Patients with any type of allergy to local anesthesia
* Patients refusing to be part of the study (refusal to sign consent)
* Any complication during surgery or anesthesia

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | within 1 week postoperatively
  The primary aim is to compare the effect of paravertebral block with general anesthesia versus general anesthesia alone on postoperative pain after laparoscopic sleeve gastrectomy surgeries. Pain will be assessed using the Visual Analogue scale (VAS) with a score of 0 denoting no pain and 10 maximum possible pain.

SECONDARY OUTCOMES:
ambulation | within 1 week postoperatively
  The secondary aim is to assess the time of first movement (early ambulation) between both groups. This will be assessed via a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Saleh Kanawati, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon